CLINICAL TRIAL: NCT01148329
Title: PROMUS™ Element™ Everolimus-Eluting Coronary Stent System European Post- Approval Surveillance Study To Evaluate Real World Clinical Outcomes Data for the PROMUS™ Element™ Coronary Stent System in Unselected Patients in Routine Clinical Practice
Brief Title: PROMUS™ Element™ Everolimus-Eluting Coronary Stent System European Post-Approval Surveillance Study
Acronym: PE-Prove
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Pharmaceutical Research Associates (Other); Medidata Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: S2057
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Coronary Heart Disease
Keywords: Coronary stenting; Drug-eluting stent; Post-market surveillance study; Promus Element stent
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single arm observational study: To evaluate real world clinical outcomes data for the PROMUS™ Element™ Coronary Stent System in unselected patients in routine clinical practice
  Interventions: Device: Coronary stenting

INTERVENTIONS:
Device: Coronary stenting — The PROMUS™ Element™ Everolimus Eluting Coronary Stent System is indicated for improving coronary luminal diameter in patients with symptomatic ischemic heart disease due to discrete de novo native coronary artery lesions. The treated lesion length should be less than the nominal stent length (8 mm, 12 mm, 16 mm, 20 mm, 24 mm, 28 mm, 32 mm, 38mm) with a reference vessel diameter of 2.25 mm - 4.0 mm.

SUMMARY:
The goal of the PROMUS™ Element™ Everolimus-Eluting Coronary Stent System European Post- Approval Surveillance Study is to evaluate real world clinical outcomes data for the PROMUS™ Element™ Coronary Stent System in unselected patients in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* According to Instructions For Use

Exclusion Criteria:

* Contraindications according to Instructions for Use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are candidates for Coronary artery stenting, signed the Informed Consent Form and are eligible to receive a PROMUS™ Element™ stent will be evaluated for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1010 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | One year
  Overall and PROMUS™ Element™ stent related TVF rate (cardiac death, myocardial infarction (MI) related to target vessel and target vessel re-intervention (TVR)) at 12 months post stent implantation.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) rates (cardiac death, MI, TVR) | 30 days, 6 months, 12 months and then annually through 5 years
  Overall and PROMUS™ Element™ stent-related MACE rates (cardiac death, MI, TVR).
Death or MI rates | 30 days, 6 months, 12 months and then annually through 5 years
  Overall and PROMUS™ Element™ stent-related cardiac death or MI rates
TVR rates | 30 days, 6 months, 12 months and then annually through 5 years
  Overall and PROMUS™ Element™ stent-related TVR rates.
Cardiac death rates | 30 days, 6 months, 12 months and then annually through 5 years
  Overall and PROMUS™ Element™ stent-related cardiac death rates.
MI Rates | 30 days, 6 months, 12 months and then annually through 5 years
  Overall and PROMUS™ Element™ stent-related MI rates.
All death rates | 30 days, 6 months, 12 months and then annually through 5 years
  All death rates
Non-cardiac death rates | 30 days, 6 months, 12 months and then annually through 5 years
  Non-cardiac death rates
All death or MI rates | 30 days, 6 months, 12 months and then annually through 5 years
  All death and MI rates

CONTACTS AND LOCATIONS:
Overall Officials: Raul Moreno, MD PhD, Principal Investigator — Hospital La Paz, Spain; Peter Maurer, PhD, Study Director — Boston Scientific Corporation
Locations (40):
- Austria (3):
  - Allgemeines Krankenhaus der Stadt Linz, Linz
  - Medizinische Universität Wien, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (2):
  - Virga Jesse Ziekenhuis, Hasselt
  - Centre Hôpital Universitaire Sart Tilman, Liège
- Denmark (2):
  - Odense University Hospital, Odense
  - Roskilde Sygehus, Roskilde
- France (6):
  - Centre Hospitalier Privé Saint Martin gds, Caen
  - Le Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Polyclinique les Fleurs, Ollioules
  - Clinique St. Martin, Pessac
  - Clinique Saint-Hilaire Rouen, Rouen
  - Clinique Pasteur, Toulouse
- Germany (8):
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Klinikum Leverkusen, Leverkusen, North Rhine-Westphalia
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Herz-Kreislauf-Zentrum Segeberger Kliniken GmbH, Bad Segeberg
  - Klinikum Darmstadt, Darmstadt
  - Med. Hochschule Hannover, Hanover
  - Schwarzwald Baar Klinikum Villingen-Schwenningen, Villingen-Schwenningen
- Dept. of Internal Medicine and Cardiological Center, Szeged, Hungary
- Ireland (4):
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Galway University Hospital, Galway
- Italy (4):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Centro Cardiologico Monzino, Milan
  - Clinica Mediterranea, Napoli
  - IRCCS Policlinico S. Matteo, Pavia
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario La Paz, Madrid
- United Kingdom (5):
  - Papworth Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - St. Thomas Hospital, London
  - King's College Hospital London, London
  - Freeman, Newcastle-Upon-Tyne, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No
Data are presented at the 2013 EuroPCR congress.

REFERENCES:
- [Result] Thomas MR, Birkemeyer R, Schwimmbeck P, Legrand V, Moreno R, Briguori C, Werner N, Bramucci E, Ungi I, Richardt G, Underwood PL, Dawkins KD. One-year outcomes in 1,010 unselected patients treated with the PROMUS Element everolimus-eluting stent: the multicentre PROMUS Element European Post-Approval Surveillance Study. EuroIntervention. 2015 Mar;10(11):1267-71. doi: 10.4244/EIJY15M01_07. PMID 25631367